CLINICAL TRIAL: NCT03869554
Title: Evaluation of a Screening Strategy of Fabry Disease in Patient With Renal Biopsy: Histo-Fab Study
Brief Title: Evaluation of a Screening Strategy of Fabry Disease in Patient With Renal Biopsy
Acronym: HISTOFAB
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 49RC19_0032
Record Dates: First submitted 2019-03-07; First posted 2019-03-11 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Renal Disease
MeSH Terms: conditions — Kidney Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Renal disease (Experimental): detection of Fabry disease
  Interventions: Diagnostic Test: Detection of Fabry disease

INTERVENTIONS:
Diagnostic Test: Detection of Fabry disease — Systematic detection of Fabry disease

SUMMARY:
Fabry disease is genetic X linked disease, with annual incidence of 1 in 100,000 that is certainly underestimate the true prevalence of the disease.

Renal biopsy in some patients does not allow determining the etiology of nephropathy. It is why investigators would like to evaluate the screening of Fabry patients from renal biopsy in patient with idiopathic nephropathy.

Investigator hypothesize to detect one or more cases of patients with Fabry disease in local idiopathic nephropathy population with renal biopsy.

That would allow reviewing and optimizing the target screening for Fabry Disease. The purpose would be to detect Fabry disease systematically in patients presenting a nephropathy of undetermined etiology in spite of the renal biopsy or presenting nonspecific histological characteristics.

In Fabry disease with renal impairment, proteinuria is the first sign, usually occurring in the second decade. The evolution is progressively towards end-stage renal failure during the fourth decade. The presence of renal impairment is globally associated with a poor prognosis.

Renal histology can be used to diagnose Fabry disease by revealing sphingolipid deposits identified by optical microscopy in the form of vacuoles in podocytes, distal tubule epithelial cells or in the media of the distal tubules. vascular walls. Resin inclusion with Toluidine blue staining is the staining of choice for visualizing lipid inclusions. However, this staining is not used as a first intention in routine. On the paraffin-fixed tissues, the vacuoles are less visible because they dissolve.

Thus, the renal histological analysis sometimes reveals only non-specific damage to the various structures of the kidney and may not allow identification of very evocative inclusions. Under the effect of oxidative stress induced by sphingolipid deposits, lesions of tubulo-interstitial fibrosis settle quite early. At the level of the glomerulus, glycosphingolipids lead to the production of angiotensin II and TGF-β leading to an excess production of constituents of the glomerular basement membrane inducing its thickening and glomerulosclerosis. Arteries of all sizes are also the seat of intimal thickening and media accelerating the process of intrarenal ischemia. These lesions, which may appear isolated or synchronous, and nonspecific, are sometimes in the foreground and do not point in the first line to the etiological diagnosis of Fabry disease.

Also, among the patients presenting a nephropathy of undetermined etiology in spite of the renal biopsy or presenting nonspecific histological characteristics, investigator propose to systematically detect the Fabry disease. Screening will be done in a selected population of renal biopsy patients using the dried blood spot kits.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (> 18 years old)
* Obtaining consent to participate in the study
* Patients whose clinical presentation meets at least one of the following criteria:

  * Undetermined nephropathy despite renal biopsy,
  * Nephroangiosclerosis as the predominant lesion
  * Chronic tubulointerstitial nephropathy,
  * Glomerulosclerosis,
  * Segmental and focal hyalinosis.
  * Optically normal kidney or seat of minimal lesions

Exclusion Criteria:

* Patient who has already been screened for Fabry Disease
* At least one of the following criteria:

  * Nephrotic syndrome and/or Glomerular nephropathy
  * Histological diagnosis of certain nephropathies (specific kidney lesions)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-02-03 (Actual); Primary Completion 2025-06-02 (Estimated); Study Completion 2025-08-02 (Estimated)

PRIMARY OUTCOMES:
Assess the value of screening for Fabry's disease in patients with kidney disease whose etiology remains undetermined after renal biopsy | 1 month
  number of patients diagnosed with Fabry's disease identified

SECONDARY OUTCOMES:
Estimate the prevalence of Fabry disease | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Angers, Angers, France